CLINICAL TRIAL: NCT06752668
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ORX750 in Subjects With Narcolepsy and Idiopathic Hypersomnia (CRYSTAL-1)
Brief Title: A Study of ORX750 in Participants With Narcolepsy and Idiopathic Hypersomnia
Acronym: CRYSTAL-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centessa Pharmaceuticals (UK) Limited (Industry)
Responsible Party: Sponsor
Organization: Centessa Pharmaceuticals plc (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORX750-0201; 2024-518929-15-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Narcolepsy Type 1; Narcolepsy Type 2; Idiopathic Hypersomnia
MeSH Terms: conditions — Idiopathic Hypersomnia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Narcolepsy Type 1: ORX750 and Placebo (Experimental)
  Interventions: Drug: ORX750; Drug: Placebo
- Narcolepsy Type 2: ORX750 and Placebo (Experimental)
  Interventions: Drug: ORX750; Drug: Placebo
- Idiopathic Hypersomnia: ORX750 and Placebo (Experimental)
  Interventions: Drug: ORX750; Drug: Placebo

INTERVENTIONS:
Drug: ORX750 — ORX750 capsule.
Drug: Placebo — ORX750 matching placebo capsule.

SUMMARY:
Narcolepsy Type 1 (NT1), Narcolepsy Type 2 (NT2), and Idiopathic Hypersomnia (IH) are rare conditions that make people feel very sleepy during the day (often referred to as excessive daytime sleepiness [EDS]). People living with these conditions might find it hard to stay alert and pay attention when they are at school, working, driving, or performing other daily activities.

While all conditions result in feeling sleepy, there are some differences in other common symptoms:

* NT1: People with NT1 often feel very tired during the day and experience cataplexy. Cataplexy is a sudden loss of muscle strength, which can cause someone to collapse or lose control of their muscles for a short time. This is often triggered by strong emotions, such as laughter or surprise. They may also have trouble sleeping well at night.
* NT2: People with NT2 feel sleepy during the day, just like NT1, but they do not have cataplexy.
* IH: People with IH feel tired during the day, even after sleeping a lot at night. They may sleep for long periods, take long naps, and find it hard to wake up.

Orexin is a protein in the brain that helps coordinate a system that plays an important role in helping people to stay awake during the daytime. ORX750 is designed to mimic the action of orexin. The purpose of this study is to see how safe and tolerable ORX750 is in NT1, NT2, and IH, and learn about what the drug does to the body. Another goal of the study is to see if ORX750 can help people with NT1, NT2, and IH feel less sleepy and make other symptoms better.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* BMI ≥17 and ≤37 kg/m2
* Meets the diagnostic criteria of Narcolepsy Type 1 (NT1), Type 2 (NT2) or Idiopathic Hypersomnia (IH) according to ICSD-3-TR criteria
* Is willing and able to discontinue all medications used for the treatment of narcolepsy or idiopathic hypersomnia
* Is willing and able to adhere to additional protocol requirements

Exclusion Criteria:

* A medical disorder other than NT1, NT2, or IH that is associated with excessive daytime sleepiness (EDS).
* Presence of significant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, hematological, malignancy, endocrine, neurological or psychiatric disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs | Up to Day 49
Number of Participants With Abnormal Changes From Baseline in Laboratory Tests | Up to Day 49
Number of Participants With Abnormal Change From Baseline in Vital Signs | Up to Day 49
Number of Participants With Abnormal Change From Baseline in Electrocardiograms (ECG) | Up to Day 49
Number of Participants With Suicidal Ideation or Suicidal Behavior as Measured Using Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to Day 49

SECONDARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for ORX750 | Day 1
Tmax: Time of Maximum Concentration for ORX750 | Days 1, 14 and 28
AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for ORX750 | Day 1
Cmax,ss: Maximum Observed Concentration at Steady State for ORX750 | Days 14 and 28
AUCτ: Area Under the Concentration-time Curve During a Dosing Interval at Steady State for ORX750 | Days 14 and 28
Mean sleep latency (average of the first 4 trials) in the Maintenance of Wakefulness Test (MWT) for ORX750 versus placebo. | Baseline up to Day 42
  Mean sleep latency is determined by averaging the time to falling asleep across trials
Change From Baseline in Epworth Sleepiness Scale (ESS) | Baseline up to Day 41

CONTACTS AND LOCATIONS:
Locations (27):
- United States (26):
  - Auburn, Alabama, Auburn, Alabama
  - Chandler, Arizona, Chandler, Arizona
  - Scottsdale, Arizona, Scottsdale, Arizona
  - Long Beach, California, Long Beach, California
  - Santa Ana, California, Santa Ana, California
  - Brandon, Florida, Brandon, Florida
  - Miami, Florida, Miami, Florida
  - Orlando, FL, Orlando, Florida
  - Winter Park, Florida, Winter Park, Florida
  - Atlanta, Georgia, Atlanta, Georgia
  - Riverdale, Georgia, Riverdale, Georgia
  - New Orleans, Louisiana, New Orleans, Louisiana
  - Newton, Massachusetts, Newton, Massachusetts
  - Southfield, Michigan, Southfield, Michigan
  - Sterling Heights, Michigan, Sterling Heights, Michigan
  - Henderson, Nevada, Henderson, Nevada
  - Denver, North Carolina, Denver, North Carolina
  - Huntersville, North Carolina, Huntersville, North Carolina
  - Cincinnati, Ohio, Cincinnati, Ohio
  - Cleveland, OH, Cleveland, Ohio
  - Dublin, Ohio, Dublin, Ohio
  - Willow Grove, Pennsylvania, Willow Grove, Pennsylvania
  - Columbia, South Carolina, Columbia, South Carolina
  - North Charleston, South Carolina, North Charleston, South Carolina
  - Austin, Texas, Austin, Texas
  - San Antonio, Texas, San Antonio, Texas
- Toronto, Ontario, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No